CLINICAL TRIAL: NCT01546363
Title: Tissue and Plasma Biomarkers of Lymph Node Involvement in Cervical Cancer
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: GYNCVX0002; SU-03012012-9208 (Other: Stanford University); 23080 (Other: Stanford IRB)
Record Dates: First submitted 2012-03-01; First posted 2012-03-07 (Estimated); Last update posted 2020-10-05 (Actual); Status verified 2020-10

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Tissue
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Validation
  Interventions: Other: Blood draw
- Testing
  Interventions: Other: Blood draw

INTERVENTIONS:
Other: Blood draw — phlebotomy

SUMMARY:
The purpose of this study is to measure the levels of serum proteins and other biomarkers in cervical cancer patients. We believe that some of these markers may be useful in selecting patients for specific types of cancer therapies. These markers may also help to predict response to therapy, relapse after therapy, and survival after therapy.

DETAILED DESCRIPTION:
SPECIFIC STUDY AIMS

Specific Aim 1: To use gene expression analysis of primary cervical cancers to identify a gene expression signature that predicts for lymph node metastases in this disease.

Specific Aim 2: To predict lymph node metastases by performing multiplex measurements of cancer-associated proteins and cytokines using proximity ligation assay (PLA) on plasma samples.

Specific Aim 3: To measure circulating human papilloma virus (HPV) DNA in the plasma samples of cervical cancer patients using real-time quantitative polymerase chain reaction (qPCR) and determine its ability to predict for nodal metastases.

Specific Aim 4: To use deep sequencing to evaluate gene and sequence differences between cervical cancer patients with and without lymph node metastasis.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a known or suspected cervical cancer.
* Age >=18 years.
* Patients must have no other active cancer at the time of diagnosis.
* Patients must have no history of a hysterectomy.
* Patients must be able to give informed consent.
* Patients must be willing to undergo a biopsy of the cervical tumor to provide tissue for the study.
* Patients must have completed a standard-of-care FDG-PET/CT prior to initiation of therapy, for assessment of lymph nodes.

Exclusion Criteria:

- Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Recruitment of patients for participation in this study will occur at Stanford Medical Center. All facilities are adequately equipped to meet all study requirements. Patients of this disease type are regularly treated at Stanford Cancer Center. Estimated accrual rates are based on normal patient flow.
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2012-02-24 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2020-06-29 (Actual)

PRIMARY OUTCOMES:
Biomarkers (genes and proteins) of lymph node involvement | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Kidd, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No